CLINICAL TRIAL: NCT06215040
Title: Multicenter Prospective Study for Efficacy of Asymptomatic Common Bile Duct Stone Treatment
Brief Title: The Treatment Effect for Asymptomatic Common Bile Duct Stone
Status: Recruiting | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Yeungnam University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Daegu Catholic University Medical Center (Other); Kyungpook National University Chilgok Hospital (Other); Daegu Fatima Hospital (Other)
Responsible Party: Principal Investigator, Jun Heo, Assistant Professor, Kyungpook National University Hospital
Other Study IDs: KNUH2023-09-029-001
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Choledocholithiasis; Asymptomatic Condition; Quality of Life
MeSH Terms: conditions — Choledocholithiasis; Asymptomatic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic common bile duct stone
  Interventions: Procedure: Endoscopic retrograde cholangiopancratography

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancratography — common bile duct stone removal
  Other Names: observation

SUMMARY:
This study is prospective, multicenter study for identify the characteristics of asymptomatic common bile duct stones and effectiveness of treatment.

DETAILED DESCRIPTION:
There is no conflcts for treatment of symptomatic common bile duct stone. As more imaging examination such as healthy screening, more asymptomatic common bile duct stone patients are found. Current guideline for aymptomatic common bile duct stone is removal using endoscopic retrograde cholangiopancreatography. However, the previous studies that support this guideline included patients who just underwent cholecystectomy and were diagnosed as common bile duct stone. There is no prospective study for identify the treatment effectiveness of common bile duct stone removal in asymptomatic patients who are dignosed in healthy screening. Therefore, we are going to find the effectiveness of common bile duct stone removal by comparing questionnarie before and after removal of common bile duct stone in asymptomatic and incidentally found common bile duct stone patients. In addition, we are going to follow up patients who do not want to undergo common bile duct stone removal and find the rate of cholangitis risk. We also want to identify extact complication rate for endoscopic retrograde pancreatocholangiographic procedures in asymptomatic common bile duct stone.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as common bile duct stone by image modality examination
* agreement for this study enrollment

Exclusion Criteria:

* no definite common bile duct stone by image modality examination
* symptomatic patients who complain with fever/abdominal pain that compatible with common bile duct stone related symptom
* previously diagnosed as pancreatobiliary malignancy
* previously treated by endoscopic or percutaneous treatment for bile duct stones
* severe cardio or pulmonary disease
* pregnancy or possibility of pregnancy
* who do not agree with study enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who have common bile duct stones without cholangitis symptom
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Score of quality of life | 3 months
  Compare the quality of life before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, Gyungsangbok-do, South Korea